CLINICAL TRIAL: NCT01401322
Title: Single Agent Lenalidomide in Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Single Agent Lenalidomide in Adult Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Bruno C. Medeiros, Assistant Professor of Medicine (Hematology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19607; SU-01142011-7364 (Other: Stanford University); RV_ALL_PI_0616 (Other: Celgene Corporation); HEMALL0006 (Other: OnCore)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Leukemia; Relapsed Adult Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide 50 mg/day x 28 days (Experimental): Lenalidomide 50 mg daily for 28 consecutive days every 42 days (+/-7 days). Treatment to continue until evidence of disease progression or development of unexpected toxicities not reversed by dose reductions and/or interruptions.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — 50 mg; po
  Other Names: Revlimid

SUMMARY:
Time-to-Progression (TTP)

DETAILED DESCRIPTION:
Determine the time-to-progression (TTP) for subjects with relapsed/refractory acute lymphoblastic leukemia (ALL) receiving single agent lenalidomide 50 mg/day for 28 days/cycle.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory acute lymphoblastic leukemia (ALL) with > 10% bone marrow or peripheral blood blasts per WHO-criteria. Refractory define as failure to achieve CR after prior therapy.
* Previously untreated patients > 60, if not candidates for standard induction
* Age ≥ 18
* Not a candidate for curative treatment regimens
* Unwilling or unable to receive conventional chemotherapy
* ECOG performance status ≤ 2
* Life expectancy > 2 months
* Registered to in RevAssist restricted distribution program, and willing and able to comply with the program requirement
* Females of childbearing potential (FCBP):

  * Must have a negative serum or urine pregnancy test (sensitivity of at least 50 mIU/mL) 10 to 14 days prior to study enrollment and within 24 hours prior to prescribing lenalidomide
  * Must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control
  * Agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP
* Able to adhere to the study visit schedule and other protocol requirements
* Willing and able to understand and voluntarily sign a written informed consent

Exclusion Criteria:

* Prior therapy with lenalidomide
* History of intolerance to thalidomide including development of erythema nodosum while taking thalidomide or similar drugs
* Advanced malignant hepatic tumors.
* Concomitant treatment with other anti-neoplastic agents (exception hydroxyurea)
* Anti-neoplastic treatment less than 4 weeks prior to enrollment (exception hydroxyurea)
* Use of any other experimental drug or therapy within 14 days of baseline
* Inability to swallow or absorb drug
* Active opportunistic infection or treatment for opportunistic infection within 4 weeks of first dose of study drug
* New York Heart Association Class III or IV heart failure
* Unstable angina pectoris
* Cardiac arrhythmias with rapid ventricular response (heart rate > 100 beats/minute)
* Uncontrolled psychiatric illness that would limit compliance with requirements
* Known HIV infection
* Known active hepatitis B virus (HBV) (exception seropositivity due to HBV vaccine not considered active HBV)
* Known hepatitis C virus (HCV) infection
* Pregnant
* Lactating females must agree not to breastfeed while taking lenalidomide
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation
* Creatinine ≥ 1.5 mg/dL
* Creatinine clearance ≤ 60 mL/min.
* Total bilirubin > 1.5 x institutional upper limit of normal (ULN) (exception documented Gilbert's syndrome)
* AST and ALT > 3 x institutional ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Carneiro de Medeiros, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenalidomide 50 mg/Day x 28 Days
Started | 5
Completed | 3
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Relapsed or refractory ALL (at least 1 failed prior treatment regimen)
Arm/Group | Lenalidomide 50 mg/Day x 28 Days
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 39.7 [32.4 to 69.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Progression (TTP)
Time Frame: 12 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Lenalidomide 50 mg/Day x 28 Days
Number analyzed (Participants) | 3
Days | 20 [19 to 21]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lenalidomide 50 mg/Day x 28 Days
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide 50 mg/Day x 28 Days (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Blood and lymphatic system disorders-Other, Pancytopenia (Blood and lymphatic system disorders) | 1 (2)
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1 (1)
Hepatobiliary disorders - Other, abnormal liver function (Hepatobiliary disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No